CLINICAL TRIAL: NCT05572086
Title: Dementia Care Challenges Among a Sample of Informal Caregivers in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Hasan, lecturer, Assiut University
Other Study IDs: Dementia care challenges
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dementia is a widespread incapacitating mental syndrome that carries a significant challenge for healthcare systems, persons with dementia, and their caregivers. The world health organization estimates that there is "more than 55 million persons live with dementia worldwide, and there are nearly 10 million new cases every year"

In Egypt there are many studies had investigated caregiver burden with chronic ill elderly as physical or psychiatric diseases; however, studies focusing on caregiving Patients With Dementia (PWD), especially the psychological aspect, has been raised just few years ago. Some focused on psychiatric comorbidities of care givers, others correlated caregivers' quality of life with dementia staging. Other research groups designed educational programs and psychosocial interventions for training informal caregivers with significant psychological burden reduction at the end of the studies , also another group focused their study on the negative emotions expressed by caregiver towards PWD. Still there are many aspects of caregiving not explored considering the financial burden, lack of formal educational resources, stigma, cultural and religious values related to caregiving.

DETAILED DESCRIPTION:
our study aims:

1. To assess challenges of dementia-related knowledge among a sample of dementia informal caregivers
2. To assess the needs of persons with dementia and their informal caregivers
3. To assess the burden of caregiving among a sample of dementia informal caregivers
4. To assess possible culturally related challenges of caregiving among a sample of dementia informal caregivers

The study will be carried out through face-to-face interview, telephone interview, and online survey from community sources, including support groups in social media, memory clinics, outpatient clinics (Geriatric medicine, neurology, or psychiatry), and social support groups of non-governmental organizations.

ELIGIBILITY:
Inclusion Criteria:

* Informal Caregivers aged 18 years or older
* Informal Caregiver in daily contact for care with the person with dementia for at least one year.

Exclusion Criteria:

* Informal caregivers who are unable or unwilling to communicate.
* Formal caregivers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: caregivers of patients with dementia from community or from patients coming to hospital for medical issues related to dementia with interview with their caregiver through face-to-face, on line, or telephone interview
Sampling Method: Non-Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of caregiver burden | one year
  By using Zarit Burden Interview